CLINICAL TRIAL: NCT01661439
Title: A Randomized Clinical Trial of Using Preconceptional Enoxaparin AND Low Dose Aspirin 81mg in Patient With Antiphospholipid Syndrome(APS)
Brief Title: Preconceptional Thromboprophylaxis in Recurrent PREGNANCY LOSSES Caused by Antiphospholipid Syndrome
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Woman's Health University Hospital, Egypt (Other)
Responsible Party: Principal Investigator, alaa eldeen mahmoud ismail, MD, Woman's Health University Hospital, Egypt
Other Study IDs: PCTRPL; preconceptional heparin in APS
Record Dates: First submitted 2012-07-25; First posted 2012-08-09 (Estimated); Last update posted 2014-06-23 (Estimated); Status verified 2012-03

CONDITIONS: Recurrent Pregnancy Losses; Positive Anti Phospholipid Syndrome
Keywords: Recurrent miscarriages; recurrent pregnancy loss; aps; anti coagulants in pregnancy
MeSH Terms: conditions — Abortion, Habitual | interventions — Heparin, Low-Molecular-Weight; Enoxaparin; Tinzaparin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Low molecular weight heparin: SC LMWH IN patients with recurrent pregnancy loss
  Interventions: Drug: low molecular weight heparin (enoxeparine)

INTERVENTIONS:
Drug: low molecular weight heparin (enoxeparine) — 1mg/kg enoxeparine SC daily from 1st day of the menstrual cycle and continue daily throughout the pregnancy after documentation of pregnancy,and stopped in absence of fetal cardiac activity.
  Other Names: clexane,innohep

SUMMARY:
Preconceptional use of low molecular weight heparin (enoxaparin) and aspirin in patient with recurrent miscarriages with positive anti phospholipid antibodies increase the implantation rate and the duration of pregnancy with low complications to the mother and the baby.

DETAILED DESCRIPTION:
Preconceptional heparin during follicular or luteal phase,improves the implantation rate by increasing the blood flow and increasing the implantation factors,also decreasing the pregnancy complication resulting from Antiphospholipid Syndrome (APS).

ELIGIBILITY:
Inclusion Criteria:

1. All women with recurrent first-trimester miscarriage and all women with one or more second-trimester miscarriage who screened before pregnancy for antiphospholipid antibodies.
2. To diagnose antiphospholipid syndrome it is mandatory that the woman has two positive tests at least 12 weeks apart for either lupus anticoagulant or anticardiolipin antibodies of immunoglobulin G and/or immunoglobulin M class present in a medium or high titre over 40 g/l or ml/l,or above the 99th percentile).

In the detection of lupus anticoagulant, the dilute Russell's viper venom time test together with a platelet neutralisation procedure is more sensitive and specific than either the activated partial thromboplastin time test or the kaolin clotting time test. Anticardiolipin antibodies are detected using a standardised enzyme linked immunosorbent assay.

Exclusion Criteria:

1. Age above forty years old .
2. Intrauterine abnormalities (as assessed by ultrasound, hysterosonography, hysterosalpingogram, or hysteroscopy).
3. Fibroids distorting uterine cavity .
4. Abnormal parental karyotype .
5. Other identifiable causes of recurrent miscarriages (tests initiated only if clinically indicated) e.g., diabetes, thyroid disease and systemic lupus erythematosus (SLE).

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: patients with recurrent pregnancy losses either two or more recurrent miscarriages or intrauterine fetal deathes after 20 weeks of gestation with positive antiphospholipid antibodies in medium to high titer in two occasions 6 weeks apart.
Sampling Method: Probability Sample
Enrollment: 316 (Estimated)
Dates: Start 2012-03; Primary Completion 2014-06 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Pregnancy continuation beyond twelve weeks gestation | ONE YEAR
  giving low molecular weight heparin (enoxaparin) and 81 mg aspirin in patients with positive anti phospholipid antibodies with history of recurrent miscarriages or intrauterine fetal deaths in the preconceptional period one month before pregnancy with follow up as regarding the clinical pregnancy rate,the rate of continuation of pregnancy beyond 28 weeks gestation and the complications related to long term use of heparin and the severity of complication of APS in comparison to the traditional use of anticoagulant after documentation of the fetal heart rate

CONTACTS AND LOCATIONS:
Locations (1):
- Women Health Hospital, Asyut, Egypt

REFERENCES:
- [Derived] Hamulyak EN, Scheres LJ, Marijnen MC, Goddijn M, Middeldorp S. Aspirin or heparin or both for improving pregnancy outcomes in women with persistent antiphospholipid antibodies and recurrent pregnancy loss. Cochrane Database Syst Rev. 2020 May 2;5(5):CD012852. doi: 10.1002/14651858.CD012852.pub2. PMID 32358837
- [Derived] Ismail AM, Hamed AH, Saso S, Abu-Elhasan AM, Abu-Elghar MM, Abdelmeged AN. Randomized controlled study of pre-conception thromboprophylaxis among patients with recurrent spontaneous abortion related to antiphospholipid syndrome. Int J Gynaecol Obstet. 2016 Feb;132(2):219-23. doi: 10.1016/j.ijgo.2015.09.004. Epub 2015 Dec 2. PMID 26810338 (Retraction: PMID 35670077 Int J Gynaecol Obstet. 2022 Aug;158(2):497)